CLINICAL TRIAL: NCT04420260
Title: Scheme of Primary Prevention of Infection by COVID-19, in Workers: Phase II Controlled Clinical Trial, to be Carried Out in Medellín-Antioquia
Brief Title: Primary Prevention of Infection by COVID-19 in Workers
Acronym: PI-Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unidad de Investigación Genética Molecular (Network)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Beatriz Aristizabal, Beatriz H Aristizabal B, MsC immunology, MsC Medical Genetics, PhD Molecular Biolgy, Scientific director of Unidad de Investigación Genética Molecular, Unidad de Investigación Genética Molecular
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UNIGEM PT-IC-02
Record Dates: First submitted 2020-05-25; First posted 2020-06-09 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: COVID
Keywords: Coronavirus Infections, Spike Glycoprotein, Functional Food, Triple Blind Clinical Study,Efficacy-Effectiveness of Interventions
MeSH Terms: conditions — Coronavirus Infections | interventions — Placebo Effect

STUDY DESIGN:
Intervention Model Description: Combination of an oropharyngeal spray and an oral immunostimulant agent for the prevention of COVID-19 infection in workers in Medellín-Antioquia. The randomized clinical trial, parallel design, triple-blind, phase II.
  Combination of an oropharyngeal spray and an oral immunostimulant agent for the prevention of COVID-19 infection in workers in Medellín-Antioquia. The randomized clinical trial, parallel design, triple-blind, phase II.
  A two-arm is stipulated, in the following manner:
  Group A: Active principle spray + Active principle emulsion. Group B: Placebo spray + Placebo emulsion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Once the participant has given its informed consent, and the research team has verified the fulfillment of the inclusion criteria, the prospect receives a text message, to be directed to the pharmaceutical service. The numbered scheme will be dispensed with the code of the intervention, following the order from the allocation listing, provided by the CTCC. The head of the pharmaceutical service will register the date and time of the first dose. He will provide indications for the use, handling, and conservation of the products. Warning signs and symptoms and instructions for communication with the research team to address any concerns the subject may have will be reviewed. He will remind the subject to avoid its damage or loss. He will give the participant instructions to return the container and surpluses of the products at the end of the trial (day 30), he will point out that they are for personal use only and that they cannot be shared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment oropharyngeal spray + immunostimulant emulsion (Experimental): Active principle oropharyngeal spray + Active principle immunostimulant taken PO.
  Interventions: Dietary Supplement: Group A: oropharygeal spray and immunostimulant emulsion
- Placebo (Placebo Comparator): Placebo oropharyngeal spray + Placebo emulsion was taken PO.
  Interventions: Dietary Supplement: Group D:Placebo oropharyngeal spray + Placebo taken PO

INTERVENTIONS:
Dietary Supplement: Group A: oropharygeal spray and immunostimulant emulsion — Intervention 1: Preparation in a liquid solution to be used for oropharyngeal spray, composed of 3 natural bioactive substances of routine use in humans, that feature homologous molecular structures to the native viral receptor.
  Intervention 2. Preparation in an emulsion functional food presentation for oral administration, that contains the 8 bioactive compounds that have demonstrated antiviral activity and modulation of the inflammatory response recognized at the moment in the immune activation against the virus.
  Other Names: BLOCKACE2 (oropharyngeal spray) + BLOCKACE2 Emulsion (Active principle immunostimulant )
  Arms: Treatment oropharyngeal spray + immunostimulant emulsion
Dietary Supplement: Group D:Placebo oropharyngeal spray + Placebo taken PO — Intervention 1: Preparation in a liquid solution to be used for oropharyngeal spray, composed of Placebo substances of routine use in humans.
  Intervention 2. Preparation in an emulsion presentation for oral administration that contains the Placebo compounds
  Other Names: Placebo+ Placebo
  Arms: Placebo

SUMMARY:
Introduction: The SARS Co-2 contagious rate is high (Ro: 2.0-3.0). The infection is aggressive with high pathogenicity. Global confinement impacts all social and economic fields of human activity. Clinical behavior exceeds the capabilities of public health care. With the initial information on the pandemic, it is estimated that 20% of health personnel in direct contact with patients can acquire the disease, despite preventive self-care. The molecular relationship of COVID-19 with the subject's ACE2 protein encourages the virus to enter the host cell, and initiates replication and the immune response, causing an imbalance generating an immunological storm of cytokines, with serious damage to the host.

Objective: It is proposed to supply a combined scheme of two compounds by oropharyngeal spray that captures the virus before entering the target cell and orally administer immunomodulatory compounds that regulate the inflammatory response released by the virus, in order to improve the antiviral response.

Methodology: A controlled, parallel design, triple-blind, phase II clinical trial will be conducted with two study groups to compare the active compounds (oropharyngeal spray and emulsion) with placebo.

Discussion: With the application of the combined scheme of two compounds, a 75% reduction in infection is expected for workers in direct contact with COVID patients.

DETAILED DESCRIPTION:
RESEARCH QUESTION: Can the oropharyngeal spray of a viral blocking compound in conjunction with the provision of an immunostimulant emulsion, reduce the infection proportion by 2/3

ACTIVE PRINCIPLE Intervention 1. BlockACE2® spray, antimicrobial and antiviral liquid solution for mouth spray, composed of 3 natural bioactive substances proven to be used in humans, which present molecular structures homologous to the native receptor of the virus. It contains binding peptides that resemble the ACE2 receptor, which bind to viral fractions, and acts as soluble scavengers of the virus at the entrance gate, upper respiratory tract, or oropharyngeal region, preventing its entry into the target cell and decreasing the amount of virus that enters the body; consequently, they reduce their ability to generate damage.

BlockACE2® Defense, food for oral administration in the form of an emulsion with 8 bioactive components that have shown modulation of the inflammatory response. Contains natural oils, Vitamin B6, Vitamin C, Vitamin E, Vitamin D3 100 SD / S, and minerals; key micronutrients that are not normally obtained through a traditional diet. These nutrients are immunostimulants with proven capacity to enhance the cellular response against viruses, anti-inflammatory, antioxidant, and chemoprotective activity, stimulating the production of interferon I; and as a whole, they prevent the generation of an excessive immune activation process, known as an "immune storm" mediated by pro-inflammatory cytokines.

Intervention 2, Placebo:

Preparations without active components in the pharmaceutical form of the above (Intervention 1 and Intervention 2). They will be presented with the same physical characteristics such as size, shape, color, taste, smell, consistency, printed signs, weight, surface finish, internal and external; in order to guarantee the principle of masking.

RESEARCH HYPOTHESIS:

In a population with community risk of COVID-19 infection, the combined use of the study interventions (the oral antimicrobial solution in Spray BlockACE2® and the food in BlockACE2® emulsion, compared to the use of Placebo, reduces the risk of COVID-19 infection expressed in a negative PCR result in those who seroconvert to IgM, and in those who seroconvert, the higher proportion will be in the mild-moderate clinical form.

PRIMARY OBJECTIVE To establish the efficacy of the combined use of BlockACE2® oropharyngeal spray, and BlockACE2® emulsion, in comparison with placebo on the reduction of the risk of infection by COVID-19, expressed in the negative result of immunoglobulins for COVID-19 (30 days from admission to the project).

Establish the safety of the products under study by evaluating the expected and unexpected adverse events that are recorded during the use phase of the intervention scheme (30 days from project entry).

SECONDARY OBJECTIVE To establish the efficacy of the combined use of BlockACE2® spray, a soluble virus scavenger compound plus ingestion of BlockACE2® emulsion, a compound that improves the defenses of the immune system, compared to placebo, on reducing the risk of infection by COVID-19 expressed in the clinical response of the disease that is defined in three variables, mild to moderate: onset of fever, myalgia, and cough without dyspnea; severe: fever, myalgia, cough and dyspnea requiring hospital care; and critical: all the above plus ventilatory assistance in ICU.

EXPLORATORY OBJECTIVES Explore the efficacy of the combined use of BlockACE2® spray, a soluble virus scavenger compound, plus the intake of BlockACE2®, an emulsion food with key micronutrients that stimulate the antiviral cellular immune response on reducing the risk of COVID-19 infection expressed in the negative result of IgG, IgM; and the reduction of the risk of symptoms such as fever, cough, dyspnea, myalgia, or ventilatory assistance in the ICU after 15 days of finishing the scheme.

FIELD OF STUDY: Workers of every department of Conconcreto Company in the city of Medellín and Girardota

INTERVENTIONS:

Intervention 1 BLOCKACE2: Two oropharyngeal sprays of the compound, every 4 hours, during the day. For the BlockACE2 emulsion will be used 20 ml during the first 5 days and after it only 10ml every day for 30 days. Dosing of the substances in intervention 1 follows the described pharmacological characteristics, that guarantee its permanence in the oral mucosa to protect the entry pathway of the virus into the organism (Oropharynx). The dosage of the oral compounds was defined according to recommendations of the WHO for the modulation of the immune response (Emulsion).

Intervention 2 PLACEBO: spray and emulsion with similar color, smell, and texture but without the natural active compounds.

In the randomization visit V1, each participant will be assigned a treatment scheme, composed of intervention 1 and intervention 2, in sufficient quantity for the duration of the study. The pharmaceutical service will dispense the code of the scheme, following a sequential order, indicated in an allocation listing of the schemes on site. Each treatment scheme is labeled with a unique code that identifies it, and it contains One (1) device for oropharyngeal spray, with a capacity for 200 applications. One (1) bottle with 360 ml (oral). In the subsequent visits, the adherence to the dispensed schemes will be verified. The frequency of use will be checked, and dosing omissions will be registered by frequency (1 dose, once a week, more than once a week).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years.
2. Health care worker in the front line of care of suspected or confirmed cases of COVID-19.
3. Negative IgM antibodies.

Exclusion Criteria:

1. Being a participant in another trial with another drug.
2. Temperature above 38ºC.
3. Having cohabited in the past 15 days with a person diagnosed with CoV-19.
4. Pregnancy.
5. Active o past smoker.
6. Known hypersensitivity to drugs or food.
7. History of respiratory disease.
8. Underlying diseases (Hypertension, cancer, diabetes, cardiovascular disease, leukopenia).
9. Signs or symptoms of CoV-19 infection: cough, dyspnea, myalgias.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Seroconversion of IgM for COVID-19. | 1 month
  Seroconversion of IgM for COVID-19. Result of positive IgM antibodies: A previously scheduled closure visit will be conducted, the trial product will be interrupted if a case is classified as severe-critical, and clinical follow up will be continued as planned. As protocols by the Health Ministry dictate, cases will be confirmed with a PCR-RT test, for the diagnosis of COVID-19. The result of the test will be requested to document the outcome.

SECONDARY OUTCOMES:
Seroconversion of IgG for COVID-19. | through study completion, 45 days
  seroconversion of IgG

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz H Aristizabal, PhD, Principal Investigator — Unidad de Investigación Genética Molecular
Locations (1):
- Beatriz Aristizabal, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yong CY, Ong HK, Yeap SK, Ho KL, Tan WS. Recent Advances in the Vaccine Development Against Middle East Respiratory Syndrome-Coronavirus. Front Microbiol. 2019 Aug 2;10:1781. doi: 10.3389/fmicb.2019.01781. eCollection 2019. PMID 31428074
- [Background] Song Z, Xu Y, Bao L, Zhang L, Yu P, Qu Y, Zhu H, Zhao W, Han Y, Qin C. From SARS to MERS, Thrusting Coronaviruses into the Spotlight. Viruses. 2019 Jan 14;11(1):59. doi: 10.3390/v11010059. PMID 30646565
- [Background] Thomas SJ, L'Azou M, Barrett AD, Jackson NA. Fast-Track Zika Vaccine Development - Is It Possible? N Engl J Med. 2016 Sep 29;375(13):1212-6. doi: 10.1056/NEJMp1609300. No abstract available. PMID 27682032
- [Background] Koch S, Pong W, Editors. The count of companies developing vaccines for coronavirus rises 2020 [Internet]. Redwood: BioCentury; 2020 [cited 2020 Feb 16]. Available from: https://www.biocentury.com/article/304412
- [Background] Ma-Lauer Y, Zheng Y, Malesevic M, von Brunn B, Fischer G, von Brunn A. Influences of cyclosporin A and non-immunosuppressive derivatives on cellular cyclophilins and viral nucleocapsid protein during human coronavirus 229E replication. Antiviral Res. 2020 Jan;173:104620. doi: 10.1016/j.antiviral.2019.104620. Epub 2019 Oct 18. PMID 31634494
- [Background] Shakya A, Bhat HR, Ghosh SK. Update on Nitazoxanide: A Multifunctional Chemotherapeutic Agent. Curr Drug Discov Technol. 2018;15(3):201-213. doi: 10.2174/1570163814666170727130003. PMID 28748751
- [Background] Pervushin K, Tan E, Parthasarathy K, Lin X, Jiang FL, Yu D, Vararattanavech A, Soong TW, Liu DX, Torres J. Structure and inhibition of the SARS coronavirus envelope protein ion channel. PLoS Pathog. 2009 Jul;5(7):e1000511. doi: 10.1371/journal.ppat.1000511. Epub 2009 Jul 10. PMID 19593379
- [Background] Barton C, Kouokam JC, Lasnik AB, Foreman O, Cambon A, Brock G, Montefiori DC, Vojdani F, McCormick AA, O'Keefe BR, Palmer KE. Activity of and effect of subcutaneous treatment with the broad-spectrum antiviral lectin griffithsin in two laboratory rodent models. Antimicrob Agents Chemother. 2014;58(1):120-7. doi: 10.1128/AAC.01407-13. Epub 2013 Oct 21. PMID 24145548
- [Background] Pruijssers AJ, Denison MR. Nucleoside analogues for the treatment of coronavirus infections. Curr Opin Virol. 2019 Apr;35:57-62. doi: 10.1016/j.coviro.2019.04.002. Epub 2019 May 21. PMID 31125806
- [Background] Totura AL, Bavari S. Broad-spectrum coronavirus antiviral drug discovery. Expert Opin Drug Discov. 2019 Apr;14(4):397-412. doi: 10.1080/17460441.2019.1581171. Epub 2019 Mar 8. PMID 30849247
- [Background] Mielech AM, Kilianski A, Baez-Santos YM, Mesecar AD, Baker SC. MERS-CoV papain-like protease has deISGylating and deubiquitinating activities. Virology. 2014 Feb;450-451:64-70. doi: 10.1016/j.virol.2013.11.040. Epub 2013 Dec 22. PMID 24503068
- [Background] Momattin H, Al-Ali AY, Al-Tawfiq JA. A Systematic Review of therapeutic agents for the treatment of the Middle East Respiratory Syndrome Coronavirus (MERS-CoV). Travel Med Infect Dis. 2019 Jul-Aug;30:9-18. doi: 10.1016/j.tmaid.2019.06.012. Epub 2019 Jun 25. PMID 31252170
- [Background] Sutton TC, Subbarao K. Development of animal models against emerging coronaviruses: From SARS to MERS coronavirus. Virology. 2015 May;479-480:247-58. doi: 10.1016/j.virol.2015.02.030. Epub 2015 Mar 16. PMID 25791336
- [Background] Mubarak A, Alturaiki W, Hemida MG. Middle East Respiratory Syndrome Coronavirus (MERS-CoV): Infection, Immunological Response, and Vaccine Development. J Immunol Res. 2019 Apr 7;2019:6491738. doi: 10.1155/2019/6491738. eCollection 2019. PMID 31089478
- [Background] Wiley JA, Richert LE, Swain SD, Harmsen A, Barnard DL, Randall TD, Jutila M, Douglas T, Broomell C, Young M, Harmsen A. Inducible bronchus-associated lymphoid tissue elicited by a protein cage nanoparticle enhances protection in mice against diverse respiratory viruses. PLoS One. 2009 Sep 23;4(9):e7142. doi: 10.1371/journal.pone.0007142. PMID 19774076
- [Background] Wohlford-Lenane CL, Meyerholz DK, Perlman S, Zhou H, Tran D, Selsted ME, McCray PB Jr. Rhesus theta-defensin prevents death in a mouse model of severe acute respiratory syndrome coronavirus pulmonary disease. J Virol. 2009 Nov;83(21):11385-90. doi: 10.1128/JVI.01363-09. Epub 2009 Aug 26. PMID 19710146
- [Background] Adedeji AO, Sarafianos SG. Antiviral drugs specific for coronaviruses in preclinical development. Curr Opin Virol. 2014 Oct;8:45-53. doi: 10.1016/j.coviro.2014.06.002. Epub 2014 Jul 2. PMID 24997250
- [Background] Al-Tawfiq JA, Hinedi K, Ghandour J, Khairalla H, Musleh S, Ujayli A, Memish ZA. Middle East respiratory syndrome coronavirus: a case-control study of hospitalized patients. Clin Infect Dis. 2014 Jul 15;59(2):160-5. doi: 10.1093/cid/ciu226. Epub 2014 Apr 9. PMID 24723278
- [Background] Baez-Santos YM, St John SE, Mesecar AD. The SARS-coronavirus papain-like protease: structure, function and inhibition by designed antiviral compounds. Antiviral Res. 2015 Mar;115:21-38. doi: 10.1016/j.antiviral.2014.12.015. Epub 2014 Dec 29. PMID 25554382
- [Background] Rider TH, Zook CE, Boettcher TL, Wick ST, Pancoast JS, Zusman BD. Broad-spectrum antiviral therapeutics. PLoS One. 2011;6(7):e22572. doi: 10.1371/journal.pone.0022572. Epub 2011 Jul 27. PMID 21818340
- [Background] Lundin A, Dijkman R, Bergstrom T, Kann N, Adamiak B, Hannoun C, Kindler E, Jonsdottir HR, Muth D, Kint J, Forlenza M, Muller MA, Drosten C, Thiel V, Trybala E. Targeting membrane-bound viral RNA synthesis reveals potent inhibition of diverse coronaviruses including the middle East respiratory syndrome virus. PLoS Pathog. 2014 May 29;10(5):e1004166. doi: 10.1371/journal.ppat.1004166. eCollection 2014 May. PMID 24874215
- [Background] Shirato K, Kawase M, Matsuyama S. Middle East respiratory syndrome coronavirus infection mediated by the transmembrane serine protease TMPRSS2. J Virol. 2013 Dec;87(23):12552-61. doi: 10.1128/JVI.01890-13. Epub 2013 Sep 11. PMID 24027332
- [Background] Millet JK, Whittaker GR. Host cell entry of Middle East respiratory syndrome coronavirus after two-step, furin-mediated activation of the spike protein. Proc Natl Acad Sci U S A. 2014 Oct 21;111(42):15214-9. doi: 10.1073/pnas.1407087111. Epub 2014 Oct 6. PMID 25288733
- [Background] Chan JF, Lau SK, To KK, Cheng VC, Woo PC, Yuen KY. Middle East respiratory syndrome coronavirus: another zoonotic betacoronavirus causing SARS-like disease. Clin Microbiol Rev. 2015 Apr;28(2):465-522. doi: 10.1128/CMR.00102-14. PMID 25810418
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Rothe C, Schunk M, Sothmann P, Bretzel G, Froeschl G, Wallrauch C, Zimmer T, Thiel V, Janke C, Guggemos W, Seilmaier M, Drosten C, Vollmar P, Zwirglmaier K, Zange S, Wolfel R, Hoelscher M. Transmission of 2019-nCoV Infection from an Asymptomatic Contact in Germany. N Engl J Med. 2020 Mar 5;382(10):970-971. doi: 10.1056/NEJMc2001468. Epub 2020 Jan 30. No abstract available. PMID 32003551
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Cheng RZ. Can early and high intravenous dose of vitamin C prevent and treat coronavirus disease 2019 (COVID-19)? Med Drug Discov. 2020 Mar;5:100028. doi: 10.1016/j.medidd.2020.100028. Epub 2020 Mar 26. No abstract available. PMID 32328576
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Killerby ME, Biggs HM, Midgley CM, Gerber SI, Watson JT. Middle East Respiratory Syndrome Coronavirus Transmission. Emerg Infect Dis. 2020 Feb;26(2):191-198. doi: 10.3201/eid2602.190697. PMID 31961300
- [Background] Sheahan TP, Sims AC, Leist SR, Schafer A, Won J, Brown AJ, Montgomery SA, Hogg A, Babusis D, Clarke MO, Spahn JE, Bauer L, Sellers S, Porter D, Feng JY, Cihlar T, Jordan R, Denison MR, Baric RS. Comparative therapeutic efficacy of remdesivir and combination lopinavir, ritonavir, and interferon beta against MERS-CoV. Nat Commun. 2020 Jan 10;11(1):222. doi: 10.1038/s41467-019-13940-6. PMID 31924756
- [Background] Hijawi B, Abdallat M, Sayaydeh A, Alqasrawi S, Haddadin A, Jaarour N, Alsheikh S, Alsanouri T. Novel coronavirus infections in Jordan, April 2012: epidemiological findings from a retrospective investigation. East Mediterr Health J. 2013;19 Suppl 1:S12-8. PMID 23888790
- [Background] de Groot RJ, Baker SC, Baric RS, Brown CS, Drosten C, Enjuanes L, Fouchier RA, Galiano M, Gorbalenya AE, Memish ZA, Perlman S, Poon LL, Snijder EJ, Stephens GM, Woo PC, Zaki AM, Zambon M, Ziebuhr J. Middle East respiratory syndrome coronavirus (MERS-CoV): announcement of the Coronavirus Study Group. J Virol. 2013 Jul;87(14):7790-2. doi: 10.1128/JVI.01244-13. Epub 2013 May 15. No abstract available. PMID 23678167
- [Background] Zhao Z, Zhang F, Xu M, Huang K, Zhong W, Cai W, Yin Z, Huang S, Deng Z, Wei M, Xiong J, Hawkey PM. Description and clinical treatment of an early outbreak of severe acute respiratory syndrome (SARS) in Guangzhou, PR China. J Med Microbiol. 2003 Aug;52(Pt 8):715-720. doi: 10.1099/jmm.0.05320-0. PMID 12867568
- [Background] Wu A, Peng Y, Huang B, Ding X, Wang X, Niu P, Meng J, Zhu Z, Zhang Z, Wang J, Sheng J, Quan L, Xia Z, Tan W, Cheng G, Jiang T. Genome Composition and Divergence of the Novel Coronavirus (2019-nCoV) Originating in China. Cell Host Microbe. 2020 Mar 11;27(3):325-328. doi: 10.1016/j.chom.2020.02.001. Epub 2020 Feb 7. PMID 32035028
- [Background] Lu R, Zhao X, Li J, Niu P, Yang B, Wu H, Wang W, Song H, Huang B, Zhu N, Bi Y, Ma X, Zhan F, Wang L, Hu T, Zhou H, Hu Z, Zhou W, Zhao L, Chen J, Meng Y, Wang J, Lin Y, Yuan J, Xie Z, Ma J, Liu WJ, Wang D, Xu W, Holmes EC, Gao GF, Wu G, Chen W, Shi W, Tan W. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Feb 22;395(10224):565-574. doi: 10.1016/S0140-6736(20)30251-8. Epub 2020 Jan 30. PMID 32007145
- [Background] Lau SKP, Zhang L, Luk HKH, Xiong L, Peng X, Li KSM, He X, Zhao PS, Fan RYY, Wong ACP, Ahmed SS, Cai JP, Chan JFW, Sun Y, Jin D, Chen H, Lau TCK, Kok RKH, Li W, Yuen KY, Woo PCY. Receptor Usage of a Novel Bat Lineage C Betacoronavirus Reveals Evolution of Middle East Respiratory Syndrome-Related Coronavirus Spike Proteins for Human Dipeptidyl Peptidase 4 Binding. J Infect Dis. 2018 Jun 20;218(2):197-207. doi: 10.1093/infdis/jiy018. PMID 29346682
- [Background] Lau SK, Li KS, Tsang AK, Lam CS, Ahmed S, Chen H, Chan KH, Woo PC, Yuen KY. Genetic characterization of Betacoronavirus lineage C viruses in bats reveals marked sequence divergence in the spike protein of pipistrellus bat coronavirus HKU5 in Japanese pipistrelle: implications for the origin of the novel Middle East respiratory syndrome coronavirus. J Virol. 2013 Aug;87(15):8638-50. doi: 10.1128/JVI.01055-13. Epub 2013 May 29. PMID 23720729
- [Background] Chu DKW, Hui KPY, Perera RAPM, Miguel E, Niemeyer D, Zhao J, Channappanavar R, Dudas G, Oladipo JO, Traore A, Fassi-Fihri O, Ali A, Demissie GF, Muth D, Chan MCW, Nicholls JM, Meyerholz DK, Kuranga SA, Mamo G, Zhou Z, So RTY, Hemida MG, Webby RJ, Roger F, Rambaut A, Poon LLM, Perlman S, Drosten C, Chevalier V, Peiris M. MERS coronaviruses from camels in Africa exhibit region-dependent genetic diversity. Proc Natl Acad Sci U S A. 2018 Mar 20;115(12):3144-3149. doi: 10.1073/pnas.1718769115. Epub 2018 Mar 5. PMID 29507189
- [Background] Paden CR, Yusof MFBM, Al Hammadi ZM, Queen K, Tao Y, Eltahir YM, Elsayed EA, Marzoug BA, Bensalah OKA, Khalafalla AI, Al Mulla M, Khudhair A, Elkheir KA, Issa ZB, Pradeep K, Elsaleh FN, Imambaccus H, Sasse J, Weber S, Shi M, Zhang J, Li Y, Pham H, Kim L, Hall AJ, Gerber SI, Al Hosani FI, Tong S, Al Muhairi SSM. Zoonotic origin and transmission of Middle East respiratory syndrome coronavirus in the UAE. Zoonoses Public Health. 2018 May;65(3):322-333. doi: 10.1111/zph.12435. Epub 2017 Dec 13. PMID 29239118
- [Background] Li W, Shi Z, Yu M, Ren W, Smith C, Epstein JH, Wang H, Crameri G, Hu Z, Zhang H, Zhang J, McEachern J, Field H, Daszak P, Eaton BT, Zhang S, Wang LF. Bats are natural reservoirs of SARS-like coronaviruses. Science. 2005 Oct 28;310(5748):676-9. doi: 10.1126/science.1118391. Epub 2005 Sep 29. PMID 16195424
- [Background] Hu B, Zeng LP, Yang XL, Ge XY, Zhang W, Li B, Xie JZ, Shen XR, Zhang YZ, Wang N, Luo DS, Zheng XS, Wang MN, Daszak P, Wang LF, Cui J, Shi ZL. Discovery of a rich gene pool of bat SARS-related coronaviruses provides new insights into the origin of SARS coronavirus. PLoS Pathog. 2017 Nov 30;13(11):e1006698. doi: 10.1371/journal.ppat.1006698. eCollection 2017 Nov. PMID 29190287
- [Background] Lau SK, Woo PC, Li KS, Huang Y, Tsoi HW, Wong BH, Wong SS, Leung SY, Chan KH, Yuen KY. Severe acute respiratory syndrome coronavirus-like virus in Chinese horseshoe bats. Proc Natl Acad Sci U S A. 2005 Sep 27;102(39):14040-5. doi: 10.1073/pnas.0506735102. Epub 2005 Sep 16. PMID 16169905
- [Background] Song HD, Tu CC, Zhang GW, Wang SY, Zheng K, Lei LC, Chen QX, Gao YW, Zhou HQ, Xiang H, Zheng HJ, Chern SW, Cheng F, Pan CM, Xuan H, Chen SJ, Luo HM, Zhou DH, Liu YF, He JF, Qin PZ, Li LH, Ren YQ, Liang WJ, Yu YD, Anderson L, Wang M, Xu RH, Wu XW, Zheng HY, Chen JD, Liang G, Gao Y, Liao M, Fang L, Jiang LY, Li H, Chen F, Di B, He LJ, Lin JY, Tong S, Kong X, Du L, Hao P, Tang H, Bernini A, Yu XJ, Spiga O, Guo ZM, Pan HY, He WZ, Manuguerra JC, Fontanet A, Danchin A, Niccolai N, Li YX, Wu CI, Zhao GP. Cross-host evolution of severe acute respiratory syndrome coronavirus in palm civet and human. Proc Natl Acad Sci U S A. 2005 Feb 15;102(7):2430-5. doi: 10.1073/pnas.0409608102. Epub 2005 Feb 4. PMID 15695582
- [Background] Wang M, Xu HF, Zhang ZB, Zou XZ, Gao Y, Liu XN, Lu EJ, Liang CY, Pan BY, Wu SJ. [Analysis on the risk factors of severe acute respiratory syndromes coronavirus infection in workers from animal markets]. Zhonghua Liu Xing Bing Xue Za Zhi. 2004 Jun;25(6):503-5. Chinese. PMID 15231128
- [Background] Forni D, Cagliani R, Clerici M, Sironi M. Molecular Evolution of Human Coronavirus Genomes. Trends Microbiol. 2017 Jan;25(1):35-48. doi: 10.1016/j.tim.2016.09.001. Epub 2016 Oct 19. PMID 27743750
- [Background] Su S, Wong G, Shi W, Liu J, Lai ACK, Zhou J, Liu W, Bi Y, Gao GF. Epidemiology, Genetic Recombination, and Pathogenesis of Coronaviruses. Trends Microbiol. 2016 Jun;24(6):490-502. doi: 10.1016/j.tim.2016.03.003. Epub 2016 Mar 21. PMID 27012512
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Ithete NL, Stoffberg S, Corman VM, Cottontail VM, Richards LR, Schoeman MC, Drosten C, Drexler JF, Preiser W. Close relative of human Middle East respiratory syndrome coronavirus in bat, South Africa. Emerg Infect Dis. 2013 Oct;19(10):1697-9. doi: 10.3201/eid1910.130946. No abstract available. PMID 24050621
- [Background] Sarris J, Kavanagh DJ. Kava and St. John's Wort: current evidence for use in mood and anxiety disorders. J Altern Complement Med. 2009 Aug;15(8):827-36. doi: 10.1089/acm.2009.0066. PMID 19614563
- [Background] Alagaili AN, Briese T, Mishra N, Kapoor V, Sameroff SC, Burbelo PD, de Wit E, Munster VJ, Hensley LE, Zalmout IS, Kapoor A, Epstein JH, Karesh WB, Daszak P, Mohammed OB, Lipkin WI. Middle East respiratory syndrome coronavirus infection in dromedary camels in Saudi Arabia. mBio. 2014 Feb 25;5(2):e00884-14. doi: 10.1128/mBio.00884-14. PMID 24570370
- [Background] Guan Y, Zheng BJ, He YQ, Liu XL, Zhuang ZX, Cheung CL, Luo SW, Li PH, Zhang LJ, Guan YJ, Butt KM, Wong KL, Chan KW, Lim W, Shortridge KF, Yuen KY, Peiris JS, Poon LL. Isolation and characterization of viruses related to the SARS coronavirus from animals in southern China. Science. 2003 Oct 10;302(5643):276-8. doi: 10.1126/science.1087139. Epub 2003 Sep 4. PMID 12958366
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Raj VS, Mou H, Smits SL, Dekkers DH, Muller MA, Dijkman R, Muth D, Demmers JA, Zaki A, Fouchier RA, Thiel V, Drosten C, Rottier PJ, Osterhaus AD, Bosch BJ, Haagmans BL. Dipeptidyl peptidase 4 is a functional receptor for the emerging human coronavirus-EMC. Nature. 2013 Mar 14;495(7440):251-4. doi: 10.1038/nature12005. PMID 23486063
- [Background] Qian Z, Travanty EA, Oko L, Edeen K, Berglund A, Wang J, Ito Y, Holmes KV, Mason RJ. Innate immune response of human alveolar type II cells infected with severe acute respiratory syndrome-coronavirus. Am J Respir Cell Mol Biol. 2013 Jun;48(6):742-8. doi: 10.1165/rcmb.2012-0339OC. PMID 23418343
- [Background] Ji W, Li X. Response to comments on "Cross-species Transmission of the Newly Identified Coronavirus 2019-nCoV" and "Codon bias analysis may be insufficient for identifying host(s) of a novel virus". J Med Virol. 2020 Sep;92(9):1440. doi: 10.1002/jmv.26048. Epub 2020 Jul 14. No abstract available. PMID 32437080
- [Background] Hui DS, I Azhar E, Madani TA, Ntoumi F, Kock R, Dar O, Ippolito G, Mchugh TD, Memish ZA, Drosten C, Zumla A, Petersen E. The continuing 2019-nCoV epidemic threat of novel coronaviruses to global health - The latest 2019 novel coronavirus outbreak in Wuhan, China. Int J Infect Dis. 2020 Feb;91:264-266. doi: 10.1016/j.ijid.2020.01.009. Epub 2020 Jan 14. No abstract available. PMID 31953166
- [Background] Chen Y, Liu Q, Guo D. Emerging coronaviruses: Genome structure, replication, and pathogenesis. J Med Virol. 2020 Apr;92(4):418-423. doi: 10.1002/jmv.25681. Epub 2020 Feb 7. PMID 31967327
- [Background] Khan S, Nabi G, Han G, Siddique R, Lian S, Shi H, Bashir N, Ali A, Shereen MA. Novel coronavirus: how things are in Wuhan. Clin Microbiol Infect. 2020 Apr;26(4):399-400. doi: 10.1016/j.cmi.2020.02.005. Epub 2020 Feb 11. No abstract available. PMID 32058086
- [Background] Zaki AM, van Boheemen S, Bestebroer TM, Osterhaus AD, Fouchier RA. Isolation of a novel coronavirus from a man with pneumonia in Saudi Arabia. N Engl J Med. 2012 Nov 8;367(19):1814-20. doi: 10.1056/NEJMoa1211721. Epub 2012 Oct 17. PMID 23075143
- [Background] Bawazir A, Al-Mazroo E, Jradi H, Ahmed A, Badri M. MERS-CoV infection: Mind the public knowledge gap. J Infect Public Health. 2018 Jan-Feb;11(1):89-93. doi: 10.1016/j.jiph.2017.05.003. Epub 2017 Jun 21. PMID 28647126
- [Background] Zhong NS, Zheng BJ, Li YM, Poon, Xie ZH, Chan KH, Li PH, Tan SY, Chang Q, Xie JP, Liu XQ, Xu J, Li DX, Yuen KY, Peiris, Guan Y. Epidemiology and cause of severe acute respiratory syndrome (SARS) in Guangdong, People's Republic of China, in February, 2003. Lancet. 2003 Oct 25;362(9393):1353-8. doi: 10.1016/s0140-6736(03)14630-2. PMID 14585636
- [Background] Cui J, Li F, Shi ZL. Origin and evolution of pathogenic coronaviruses. Nat Rev Microbiol. 2019 Mar;17(3):181-192. doi: 10.1038/s41579-018-0118-9. PMID 30531947
- [Background] Wu JT, Leung K, Leung GM. Nowcasting and forecasting the potential domestic and international spread of the 2019-nCoV outbreak originating in Wuhan, China: a modelling study. Lancet. 2020 Feb 29;395(10225):689-697. doi: 10.1016/S0140-6736(20)30260-9. Epub 2020 Jan 31. PMID 32014114
- [Background] Kim K, Andrew SA, Jung K. Public Health Network Structure and Collaboration Effectiveness during the 2015 MERS Outbreak in South Korea: An Institutional Collective Action Framework. Int J Environ Res Public Health. 2017 Sep 15;14(9):1064. doi: 10.3390/ijerph14091064. PMID 28914780
- [Background] Malave A, Elamin EM. Severe Acute Respiratory Syndrome (SARS)-Lessons for Future Pandemics. Virtual Mentor. 2010 Sep 1;12(9):719-25. doi: 10.1001/virtualmentor.2010.12.9.cprl1-1009. No abstract available. PMID 23186878
- [Background] Park JE, Jung S, Kim A, Park JE. MERS transmission and risk factors: a systematic review. BMC Public Health. 2018 May 2;18(1):574. doi: 10.1186/s12889-018-5484-8. PMID 29716568
- [Background] Al-Tawfiq JA, Auwaerter PG. Healthcare-associated infections: the hallmark of Middle East respiratory syndrome coronavirus with review of the literature. J Hosp Infect. 2019 Jan;101(1):20-29. doi: 10.1016/j.jhin.2018.05.021. Epub 2018 Jun 1. PMID 29864486
- [Background] Paules CI, Marston HD, Fauci AS. Coronavirus Infections-More Than Just the Common Cold. JAMA. 2020 Feb 25;323(8):707-708. doi: 10.1001/jama.2020.0757. No abstract available. PMID 31971553
- [Background] Arabi YM, Alothman A, Balkhy HH, Al-Dawood A, AlJohani S, Al Harbi S, Kojan S, Al Jeraisy M, Deeb AM, Assiri AM, Al-Hameed F, AlSaedi A, Mandourah Y, Almekhlafi GA, Sherbeeni NM, Elzein FE, Memon J, Taha Y, Almotairi A, Maghrabi KA, Qushmaq I, Al Bshabshe A, Kharaba A, Shalhoub S, Jose J, Fowler RA, Hayden FG, Hussein MA; And the MIRACLE trial group. Treatment of Middle East Respiratory Syndrome with a combination of lopinavir-ritonavir and interferon-beta1b (MIRACLE trial): study protocol for a randomized controlled trial. Trials. 2018 Jan 30;19(1):81. doi: 10.1186/s13063-017-2427-0. PMID 29382391
- [Background] Nassar MS, Bakhrebah MA, Meo SA, Alsuabeyl MS, Zaher WA. Middle East Respiratory Syndrome Coronavirus (MERS-CoV) infection: epidemiology, pathogenesis and clinical characteristics. Eur Rev Med Pharmacol Sci. 2018 Aug;22(15):4956-4961. doi: 10.26355/eurrev_201808_15635. PMID 30070331
- [Background] Kim KH, Tandi TE, Choi JW, Moon JM, Kim MS. Middle East respiratory syndrome coronavirus (MERS-CoV) outbreak in South Korea, 2015: epidemiology, characteristics and public health implications. J Hosp Infect. 2017 Feb;95(2):207-213. doi: 10.1016/j.jhin.2016.10.008. Epub 2016 Oct 14. PMID 28153558
- [Background] Al-Omari A, Rabaan AA, Salih S, Al-Tawfiq JA, Memish ZA. MERS coronavirus outbreak: Implications for emerging viral infections. Diagn Microbiol Infect Dis. 2019 Mar;93(3):265-285. doi: 10.1016/j.diagmicrobio.2018.10.011. Epub 2018 Oct 18. PMID 30413355
- [Background] de Araujo Lopes A, da Fonseca FN, Rocha TM, de Freitas LB, Araujo EVO, Wong DVT, Lima Junior RCP, Leal LKAM. Eugenol as a Promising Molecule for the Treatment of Dermatitis: Antioxidant and Anti-inflammatory Activities and Its Nanoformulation. Oxid Med Cell Longev. 2018 Dec 11;2018:8194849. doi: 10.1155/2018/8194849. eCollection 2018. PMID 30647816
- [Background] Bachiega TF, de Sousa JP, Bastos JK, Sforcin JM. Clove and eugenol in noncytotoxic concentrations exert immunomodulatory/anti-inflammatory action on cytokine production by murine macrophages. J Pharm Pharmacol. 2012 Apr;64(4):610-6. doi: 10.1111/j.2042-7158.2011.01440.x. Epub 2012 Feb 7. PMID 22420667
- [Background] Kim SS, Oh OJ, Min HY, Park EJ, Kim Y, Park HJ, Nam Han Y, Lee SK. Eugenol suppresses cyclooxygenase-2 expression in lipopolysaccharide-stimulated mouse macrophage RAW264.7 cells. Life Sci. 2003 Jun 6;73(3):337-48. doi: 10.1016/s0024-3205(03)00288-1. PMID 12757841
- [Background] Yogalakshmi B, Viswanathan P, Anuradha CV. Investigation of antioxidant, anti-inflammatory and DNA-protective properties of eugenol in thioacetamide-induced liver injury in rats. Toxicology. 2010 Feb 9;268(3):204-12. doi: 10.1016/j.tox.2009.12.018. Epub 2009 Dec 29. PMID 20036707
- [Background] Mnafgui K, Hajji R, Derbali F, Gammoudi A, Khabbabi G, Ellefi H, Allouche N, Kadri A, Gharsallah N. Anti-inflammatory, Antithrombotic and Cardiac Remodeling Preventive Effects of Eugenol in Isoproterenol-Induced Myocardial Infarction in Wistar Rat. Cardiovasc Toxicol. 2016 Oct;16(4):336-44. doi: 10.1007/s12012-015-9343-x. PMID 26391896
- [Background] Pan C, Dong Z. Antiasthmatic Effects of Eugenol in a Mouse Model of Allergic Asthma by Regulation of Vitamin D3 Upregulated Protein 1/NF-kappaB Pathway. Inflammation. 2015 Aug;38(4):1385-93. doi: 10.1007/s10753-015-0110-8. PMID 25588851
- [Background] Abuohashish HM, Khairy DA, Abdelsalam MM, Alsayyah A, Ahmed MM, Al-Rejaie SS. In-vivo assessment of the osteo-protective effects of eugenol in alveolar bone tissues. Biomed Pharmacother. 2018 Jan;97:1303-1310. doi: 10.1016/j.biopha.2017.11.068. Epub 2017 Dec 14. PMID 29156519
- [Background] Deepak V, Kasonga A, Kruger MC, Coetzee M. Inhibitory effects of eugenol on RANKL-induced osteoclast formation via attenuation of NF-kappaB and MAPK pathways. Connect Tissue Res. 2015 Jun;56(3):195-203. doi: 10.3109/03008207.2014.989320. Epub 2014 Dec 11. PMID 25405641
- [Background] Hussain T, Tan B, Yin Y, Blachier F, Tossou MC, Rahu N. Oxidative Stress and Inflammation: What Polyphenols Can Do for Us? Oxid Med Cell Longev. 2016;2016:7432797. doi: 10.1155/2016/7432797. Epub 2016 Sep 22. PMID 27738491
- [Background] Reuter S, Gupta SC, Chaturvedi MM, Aggarwal BB. Oxidative stress, inflammation, and cancer: how are they linked? Free Radic Biol Med. 2010 Dec 1;49(11):1603-16. doi: 10.1016/j.freeradbiomed.2010.09.006. Epub 2010 Sep 16. PMID 20840865
- [Background] Ambade A, Mandrekar P. Oxidative stress and inflammation: essential partners in alcoholic liver disease. Int J Hepatol. 2012;2012:853175. doi: 10.1155/2012/853175. Epub 2012 Mar 1. PMID 22500241
- [Background] Garcia N, Zazueta C, Aguilera-Aguirre L. Oxidative Stress and Inflammation in Cardiovascular Disease. Oxid Med Cell Longev. 2017;2017:5853238. doi: 10.1155/2017/5853238. Epub 2017 Apr 27. No abstract available. PMID 28536646
- [Background] Capasso A. Antioxidant action and therapeutic efficacy of Allium sativum L. Molecules. 2013 Jan 4;18(1):690-700. doi: 10.3390/molecules18010690. PMID 23292331
- [Background] Gu X, Wu H, Fu P. Allicin attenuates inflammation and suppresses HLA-B27 protein expression in ankylosing spondylitis mice. Biomed Res Int. 2013;2013:171573. doi: 10.1155/2013/171573. Epub 2013 Nov 13. PMID 24324956
- [Background] Ban JO, Yuk DY, Woo KS, Kim TM, Lee US, Jeong HS, Kim DJ, Chung YB, Hwang BY, Oh KW, Hong JT. Inhibition of cell growth and induction of apoptosis via inactivation of NF-kappaB by a sulfurcompound isolated from garlic in human colon cancer cells. J Pharmacol Sci. 2007 Aug;104(4):374-83. doi: 10.1254/jphs.fp0070789. PMID 17721042
- [Background] Macpherson LJ, Geierstanger BH, Viswanath V, Bandell M, Eid SR, Hwang S, Patapoutian A. The pungency of garlic: activation of TRPA1 and TRPV1 in response to allicin. Curr Biol. 2005 May 24;15(10):929-34. doi: 10.1016/j.cub.2005.04.018. PMID 15916949
- [Background] Alpers DH. Garlic and its potential for prevention of colorectal cancer and other conditions. Curr Opin Gastroenterol. 2009 Mar;25(2):116-21. doi: 10.1097/MOG.0b013e32831ef221. No abstract available. PMID 19528879
- [Background] Shen Y, Jia LN, Honma N, Hosono T, Ariga T, Seki T. Beneficial effects of cinnamon on the metabolic syndrome, inflammation, and pain, and mechanisms underlying these effects - a review. J Tradit Complement Med. 2012 Jan;2(1):27-32. doi: 10.1016/s2225-4110(16)30067-0. PMID 24716111
- [Background] Ta CA, Arnason JT. Mini Review of Phytochemicals and Plant Taxa with Activity as Microbial Biofilm and Quorum Sensing Inhibitors. Molecules. 2015 Dec 26;21(1):E29. doi: 10.3390/molecules21010029. PMID 26712734
- [Background] Anand David AV, Arulmoli R, Parasuraman S. Overviews of Biological Importance of Quercetin: A Bioactive Flavonoid. Pharmacogn Rev. 2016 Jul-Dec;10(20):84-89. doi: 10.4103/0973-7847.194044. PMID 28082789
- [Background] Senchina DS, Hallam JE, Dias AS, Perera MA. Human blood mononuclear cell in vitro cytokine response before and after two different strenuous exercise bouts in the presence of bloodroot and Echinacea extracts. Blood Cells Mol Dis. 2009 Nov-Dec;43(3):298-303. doi: 10.1016/j.bcmd.2009.08.003. Epub 2009 Sep 19. PMID 19766513
- [Background] Burger RA, Torres AR, Warren RP, Caldwell VD, Hughes BG. Echinacea-induced cytokine production by human macrophages. Int J Immunopharmacol. 1997 Jul;19(7):371-9. doi: 10.1016/s0192-0561(97)00061-1. PMID 9568541
- [Background] Ma XL, Meng M, Han LR, Li Z, Cao XH, Wang CL. Immunomodulatory activity of macromolecular polysaccharide isolated from Grifola frondosa. Chin J Nat Med. 2015 Dec;13(12):906-14. doi: 10.1016/S1875-5364(15)30096-0. PMID 26721709
- [Background] Tulk SE, Liao KC, Muruve DA, Li Y, Beck PL, MacDonald JA. Vitamin D(3) metabolites enhance the NLRP3-dependent secretion of IL-1beta from human THP-1 monocytic cells. J Cell Biochem. 2015 May;116(5):711-20. doi: 10.1002/jcb.24985. PMID 25639477
- [Background] Verway M, Bouttier M, Wang TT, Carrier M, Calderon M, An BS, Devemy E, McIntosh F, Divangahi M, Behr MA, White JH. Vitamin D induces interleukin-1beta expression: paracrine macrophage epithelial signaling controls M. tuberculosis infection. PLoS Pathog. 2013;9(6):e1003407. doi: 10.1371/journal.ppat.1003407. Epub 2013 Jun 6. PMID 23762029
- [Background] Rao Z, Chen X, Wu J, Xiao M, Zhang J, Wang B, Fang L, Zhang H, Wang X, Yang S, Chen Y. Vitamin D Receptor Inhibits NLRP3 Activation by Impeding Its BRCC3-Mediated Deubiquitination. Front Immunol. 2019 Dec 4;10:2783. doi: 10.3389/fimmu.2019.02783. eCollection 2019. PMID 31866999
- [Background] Lu L, Lu Q, Chen W, Li J, Li C, Zheng Z. Vitamin D3 Protects against Diabetic Retinopathy by Inhibiting High-Glucose-Induced Activation of the ROS/TXNIP/NLRP3 Inflammasome Pathway. J Diabetes Res. 2018 Feb 22;2018:8193523. doi: 10.1155/2018/8193523. eCollection 2018. PMID 29682582
- [Background] Ulbricht C, Basch E, Cheung L, Goldberg H, Hammerness P, Isaac R, Khalsa KP, Romm A, Rychlik I, Varghese M, Weissner W, Windsor RC, Wortley J. An evidence-based systematic review of elderberry and elderflower (Sambucus nigra) by the Natural Standard Research Collaboration. J Diet Suppl. 2014 Mar;11(1):80-120. doi: 10.3109/19390211.2013.859852. Epub 2014 Jan 10. PMID 24409980
- [Background] Chen C, Zuckerman DM, Brantley S, Sharpe M, Childress K, Hoiczyk E, Pendleton AR. Sambucus nigra extracts inhibit infectious bronchitis virus at an early point during replication. BMC Vet Res. 2014 Jan 16;10:24. doi: 10.1186/1746-6148-10-24. PMID 24433341
- [Background] Weng JR, Lin CS, Lai HC, Lin YP, Wang CY, Tsai YC, Wu KC, Huang SH, Lin CW. Antiviral activity of Sambucus FormosanaNakai ethanol extract and related phenolic acid constituents against human coronavirus NL63. Virus Res. 2019 Nov;273:197767. doi: 10.1016/j.virusres.2019.197767. Epub 2019 Sep 24. PMID 31560964
- [Background] Hemila H. Vitamin C supplementation and respiratory infections: a systematic review. Mil Med. 2004 Nov;169(11):920-5. doi: 10.7205/milmed.169.11.920. PMID 15605943
- [Background] Choe JY, Kim SK. Quercetin and Ascorbic Acid Suppress Fructose-Induced NLRP3 Inflammasome Activation by Blocking Intracellular Shuttling of TXNIP in Human Macrophage Cell Lines. Inflammation. 2017 Jun;40(3):980-994. doi: 10.1007/s10753-017-0542-4. PMID 28326454
- [Background] Dabbagh-Bazarbachi H, Clergeaud G, Quesada IM, Ortiz M, O'Sullivan CK, Fernandez-Larrea JB. Zinc ionophore activity of quercetin and epigallocatechin-gallate: from Hepa 1-6 cells to a liposome model. J Agric Food Chem. 2014 Aug 13;62(32):8085-93. doi: 10.1021/jf5014633. Epub 2014 Jul 31. PMID 25050823
- [Background] Kaihatsu K, Yamabe M, Ebara Y. Antiviral Mechanism of Action of Epigallocatechin-3-O-gallate and Its Fatty Acid Esters. Molecules. 2018 Sep 27;23(10):2475. doi: 10.3390/molecules23102475. PMID 30262731
- [Background] Wen CC, Kuo YH, Jan JT, Liang PH, Wang SY, Liu HG, Lee CK, Chang ST, Kuo CJ, Lee SS, Hou CC, Hsiao PW, Chien SC, Shyur LF, Yang NS. Specific plant terpenoids and lignoids possess potent antiviral activities against severe acute respiratory syndrome coronavirus. J Med Chem. 2007 Aug 23;50(17):4087-95. doi: 10.1021/jm070295s. Epub 2007 Jul 31. PMID 17663539
- [Background] Chen H, Lin H, Xie S, Huang B, Qian Y, Chen K, Niu Y, Shen HM, Cai J, Li P, Leng J, Yang H, Xia D, Wu Y. Myricetin inhibits NLRP3 inflammasome activation via reduction of ROS-dependent ubiquitination of ASC and promotion of ROS-independent NLRP3 ubiquitination. Toxicol Appl Pharmacol. 2019 Feb 15;365:19-29. doi: 10.1016/j.taap.2018.12.019. Epub 2018 Dec 27. PMID 30594691
- [Background] Yamagata K, Hashiguchi K, Yamamoto H, Tagami M. Dietary Apigenin Reduces Induction of LOX-1 and NLRP3 Expression, Leukocyte Adhesion, and Acetylated Low-Density Lipoprotein Uptake in Human Endothelial Cells Exposed to Trimethylamine-N-Oxide. J Cardiovasc Pharmacol. 2019 Dec;74(6):558-565. doi: 10.1097/FJC.0000000000000747. PMID 31815868
- [Background] Lim H, Min DS, Park H, Kim HP. Flavonoids interfere with NLRP3 inflammasome activation. Toxicol Appl Pharmacol. 2018 Sep 15;355:93-102. doi: 10.1016/j.taap.2018.06.022. Epub 2018 Jun 28. PMID 29960001
- [Background] Phillips JM, Gallagher T, Weiss SR. Neurovirulent Murine Coronavirus JHM.SD Uses Cellular Zinc Metalloproteases for Virus Entry and Cell-Cell Fusion. J Virol. 2017 Mar 29;91(8):e01564-16. doi: 10.1128/JVI.01564-16. Print 2017 Apr 15. PMID 28148786
- [Background] Romero JM, Grunwald B, Jang GH, Bavi PP, Jhaveri A, Masoomian M, Fischer SE, Zhang A, Denroche RE, Lungu IM, De Luca A, Bartlett JMS, Xu J, Li N, Dhaliwal S, Liang SB, Chadwick D, Vyas F, Bronsert P, Khokha R, McGaha TL, Notta F, Ohashi PS, Done SJ, O'Kane GM, Wilson JM, Knox JJ, Connor A, Wang Y, Zogopoulos G, Gallinger S. A Four-Chemokine Signature Is Associated with a T-cell-Inflamed Phenotype in Primary and Metastatic Pancreatic Cancer. Clin Cancer Res. 2020 Apr 15;26(8):1997-2010. doi: 10.1158/1078-0432.CCR-19-2803. Epub 2020 Jan 21. PMID 31964786
- [Background] Gorbachev AV, Kobayashi H, Kudo D, Tannenbaum CS, Finke JH, Shu S, Farber JM, Fairchild RL. CXC chemokine ligand 9/monokine induced by IFN-gamma production by tumor cells is critical for T cell-mediated suppression of cutaneous tumors. J Immunol. 2007 Feb 15;178(4):2278-86. doi: 10.4049/jimmunol.178.4.2278. PMID 17277133
- [Background] Prather AA, Janicki-Deverts D, Hall MH, Cohen S. Behaviorally Assessed Sleep and Susceptibility to the Common Cold. Sleep. 2015 Sep 1;38(9):1353-9. doi: 10.5665/sleep.4968. PMID 26118561
- [Background] Yan R, Zhang Y, Li Y, Xia L, Guo Y, Zhou Q. Structural basis for the recognition of SARS-CoV-2 by full-length human ACE2. Science. 2020 Mar 27;367(6485):1444-1448. doi: 10.1126/science.abb2762. Epub 2020 Mar 4. PMID 32132184
- [Background] Li G, Fan Y, Lai Y, Han T, Li Z, Zhou P, Pan P, Wang W, Hu D, Liu X, Zhang Q, Wu J. Coronavirus infections and immune responses. J Med Virol. 2020 Apr;92(4):424-432. doi: 10.1002/jmv.25685. Epub 2020 Feb 7. PMID 31981224
- [Background] He Y, Hara H, Nunez G. Mechanism and Regulation of NLRP3 Inflammasome Activation. Trends Biochem Sci. 2016 Dec;41(12):1012-1021. doi: 10.1016/j.tibs.2016.09.002. Epub 2016 Sep 23. PMID 27669650
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Sutterwala FS, Haasken S, Cassel SL. Mechanism of NLRP3 inflammasome activation. Ann N Y Acad Sci. 2014 Jun;1319(1):82-95. doi: 10.1111/nyas.12458. Epub 2014 May 19. PMID 24840700
- [Background] Vaduganathan M, Vardeny O, Michel T, McMurray JJV, Pfeffer MA, Solomon SD. Renin-Angiotensin-Aldosterone System Inhibitors in Patients with Covid-19. N Engl J Med. 2020 Apr 23;382(17):1653-1659. doi: 10.1056/NEJMsr2005760. Epub 2020 Mar 30. No abstract available. PMID 32227760
- [Background] Watanabe T, Barker TA, Berk BC. Angiotensin II and the endothelium: diverse signals and effects. Hypertension. 2005 Feb;45(2):163-9. doi: 10.1161/01.HYP.0000153321.13792.b9. Epub 2005 Jan 3. PMID 15630047
- [Background] Monteil V, Kwon H, Prado P, Hagelkruys A, Wimmer RA, Stahl M, Leopoldi A, Garreta E, Hurtado Del Pozo C, Prosper F, Romero JP, Wirnsberger G, Zhang H, Slutsky AS, Conder R, Montserrat N, Mirazimi A, Penninger JM. Inhibition of SARS-CoV-2 Infections in Engineered Human Tissues Using Clinical-Grade Soluble Human ACE2. Cell. 2020 May 14;181(4):905-913.e7. doi: 10.1016/j.cell.2020.04.004. Epub 2020 Apr 24. PMID 32333836
- [Background] Liu C, Zhou Q, Li Y, Garner LV, Watkins SP, Carter LJ, Smoot J, Gregg AC, Daniels AD, Jervey S, Albaiu D. Research and Development on Therapeutic Agents and Vaccines for COVID-19 and Related Human Coronavirus Diseases. ACS Cent Sci. 2020 Mar 25;6(3):315-331. doi: 10.1021/acscentsci.0c00272. Epub 2020 Mar 12. No abstract available. PMID 32226821
- [Background] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Jin Y, Yang H, Ji W, Wu W, Chen S, Zhang W, Duan G. Virology, Epidemiology, Pathogenesis, and Control of COVID-19. Viruses. 2020 Mar 27;12(4):372. doi: 10.3390/v12040372. PMID 32230900
- [Result] Schindewolf C, Menachery VD. Middle East Respiratory Syndrome Vaccine Candidates: Cautious Optimism. Viruses. 2019 Jan 17;11(1):74. doi: 10.3390/v11010074. PMID 30658390